CLINICAL TRIAL: NCT00002175
Title: Epicutaneous 1-Chloro-2, 4-Dinitrobenzene (DNCB) Patch in HIV Infection.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Honolulu Medical Group (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 265A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-01

CONDITIONS: HIV Infections
Keywords: Cohort Studies; RNA, Viral; Administration, Cutaneous; Anti-HIV Agents; Dinitrobenzenes
MeSH Terms: conditions — HIV Infections | interventions — Dinitrochlorobenzene

INTERVENTIONS:
Drug: Dinitrochlorobenzene

SUMMARY:
To evaluate the efficacy of dinitrochlorobenzene (DNCB) in patients with early HIV infection by monitoring immunologic parameters and serum HIV RNA. To facilitate the understanding of possible alterations in the immunological status of the HIV+ patient cohort.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* EITHER HIV negative or documented HIV+ by both the ELISA and Western blot tests.

For HIV+ patients:

* Patients must fail to meet the AIDS-defining criteria.
* CD4 lymphocyte count between 200 - 500 cells/mm3.

Exclusion Criteria

Co-existing Condition:

Excluded:

Patients with obvious ultra violet(UV)-irradiated skin damage in the treatment sites.

Concurrent Medication:

Excluded:

* Patients who are likely to commence antiretrovirals within the 6-month study period.
* Patients using other immunomodulator therapies or other alternative therapies.
* Patients likely to require chemotherapy during the course of the study.

Concurrent Treatment:

Excluded:

* Patients who are likely to require significant UV light exposure during the study period.
* Patients who are likely to require radiation therapy during the course of the study.

Prior Medication:

Excluded:

* Prior exposure to DNCB.
* Patients who have used antiretroviral medications within the previous 3 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Emma Clinics / The Queen's Med Ctr, Honolulu, Hawaii, United States